CLINICAL TRIAL: NCT01935804
Title: Phase 1 Study of Pioglitazone Versus Metformin on Bone Health in Postmenopausal Women With Type 2 Diabetes
Brief Title: Effect of Pioglitazone Versus Metformin on Bone Health in Postmenopausal Women With Type 2 Diabetes
Acronym: Pioglitazone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Mohammed-Salleh M. Ardawi, Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEOR-01-08
Record Dates: First submitted 2013-08-27; First posted 2013-09-05 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders
Keywords: pioglitazone; metformin; hyperglycemic agents; physiological effects of drugs; bone health
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: 1 (Experimental): Pioglitazone given 30mg/once daily for 12 months.
  Interventions: Drug: Pioglitazone
- Active comparator: 2 (Active Comparator): Metformin given 850 mg/twice daily for 12 months.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Pioglitazone — 30 mg/daily for 12 months
  Other Names: Actos
  Arms: Experimental: 1
Drug: Metformin — 850 mg/daily for 12 months
  Other Names: Glucophage
  Arms: Active comparator: 2

SUMMARY:
The study tests whether pioglitazone (PIO)as compared to metformin (MET)affects bone health including bone mineral density, bone turnover markers, and osteocyte biomarker in patients with type 2 diabetes (T2DM).

DETAILED DESCRIPTION:
Women with T2DM exhibit normal or higher bone mineral density (BMD) for their age, but with approximately twice the overall risk of bone fragility compared with nondiabetic subjects. Known the apparent association between T2DM and the risk of bone fragility, examining the effects of commonly used oral antidiabetic agents; such as MET and thiazolidinediones (TZDs; for example rosiglitazone [ROS] or PIO), on BMD and/or bone turnover is of great clinical relevance for both diabetic patients and their treating physicians. Recent clinical trials, showed that women treated with ROS had higher risk of bone fragility and self-reported adverse events. Similarly, women on long-term treatment with PIO for T2DM experienced higher incidence of distal extremity fractures. TZDs are agonists of the nuclear transcription factor peroxisome proliferator- activated receptor-γ (PPAR-γ) which increase insulin sensitivity and improve glycemic control in T2DM. PPAR (γ) acts also as a molecular factor that favours adipogenesis over osteoblastogenesis of mesenchymal stem cells. The latter was suggested as a potential mechanism for the effects of TZDs on bone among others. In humans, TZDs decrease BMD and increase bone fragility risk. This study tests whether pioglitazone as compared to MET (both are commonly used in the treatment of T2DM in Saudi Arabia and other countries) affects bone health including bone mineral density, bone turnover markers, and osteocyte biomarker in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* BMD T-score greater than -2.5 at the total hip, femoral neck, and lumbar spine;
* No prior antidiabetic therapy;
* Drug-naïve with glycosylated hemoglobin A1c (HbA1c) ≥ 7.0 to ≤ 10.0%. 53.2 mmol/mol to 88.2 mmol/mol);
* Body-mass index of 40 Kg/m2 and less;
* Stable body weight for at least 4 months.

Exclusion Criteria:

* Type 1 diabetes mellitus (presence of GAD auto antibodies);
* History of diabetes or uncontrolled hypertension;
* Treatment with antidiabetic agents including TZDs;
* Chronic diseases known to affect bone;
* Previous treatment with estrogens and other medications known to affect bone ;
* Creatinine clearance less than 60 ml/min

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in mean percentage change in BMD at various sites by Dual energy X-ray absorptiometry(DXA) from baseline and at 6, 12 months in PIO versus MET treatment group. | 6-18 months
  The primary endpoint was change in mean percentage change in BMD values at the lumbar spine (L1-L4), femoral neck and total hip by DXA from baseline and at 6 and 12 months in the PIO and the MET treatment groups.

SECONDARY OUTCOMES:
Bone turnover Markers and other Biomarkers | 6-18 months
  Secondary end-points were changes in serum sclerostin, serum bone-specific alkaline phosphatase (BSAP), serum procollagen type1 N-terminal propeptide (P1NP) and serum C-terminal crosslinking telopeptide of type 1 collagen (CTX); and urinary N-terminal crosslinking telopeptide type 1 collagen (u-NTX); serum calcium, 25-hydroxyvitamin D (25-OHD), and serum Dickkopf-1( DKK-1) at various time intervals from baseline between PIO vs MET treatment.

OTHER OUTCOMES:
Exploratory and Safety Outcomes | 6-18 months
  Other endpoints were changes in inflammatory markers (hs-CRP)
Exploratory Outcomes: lipid profile | 6-18 months
  lipid profile (total cholesterol, HDL-c, LDL-c and triglycerides)
Exploratory outcomes: liver and renal function tests | 6-18 months
  liver function tests [albumin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP)]; renal function tests (creatinine, urea, uric acid) and parathyroid hormone (PTH).
Exploratory outcomes: glycemic control | 6-18 months
  within and between treatment group comparisons of change from baseline at specified time points in HbA1c, fasting plasma glucose (FPG), fasting plasma insulin, and insulin sensitivity measured by the homeostasis model assessment (HOMA-s).
Exploratory and safety outcomes | 6-18 months
  Safety endpoints were adverse events (AEs), clinical laboratory assessments, vital signs, and electrocardiograms

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed-Salleh M Ardawi, PhD, FRCPath, Principal Investigator — Center of Excellence for Osteoporosis Research and Faculty of Medicine, King Abdulaziz University; Abdulrahim A Rouzi, FRCPC, Study Director — Center of Excellence for Osteoporosis Research, and Faculty of Medicine, King Abdulaziz University
Locations (1):
- Center of Excellence for Osteoporosis Research, King Abdulaziz University, Jeddah, Mecca Region, Saudi Arabia